CLINICAL TRIAL: NCT05724940
Title: Comparison of Clinical and Serological Differences Among Juvenile, Adult, and Late-onset Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Hemdan, assistant lecture, Sohag University
Other Study IDs: soh-med-22-12-15
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

INTERVENTIONS:
Other: clinical and serological differences among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients — All patients will be subjected to the following:
  1. Thorough medical history of the patients
  2. Full clinical examination including:
     1. General examination and vital signs.
     2. Complete rheumatological examination.
     3. SLE disease activity index SLEDAI (ref).
     4. SLICC( Systemic Lupus International Collaborating Clinics) damage index (ref).
  3. Routine investigations (complete blood picture, erythrocyte sedimentation rate and liver functions).
  4. Renal investigations:
     1. Kidney functions
     2. Urine analysis
     3. 24 hours protein in urine and/or A/C ratio
     4. Renal biopsy if indicated.
  5. ANA (Antinuclear Antibodies)test.
  6. ANA profile for the most common 19 autoantibodies by immunoblot.

SUMMARY:
Systemic lupus erythematosus (SLE) is a heterogeneous autoimmune disease with a highly variable presentation and course. It can affect virtually every organ of the body and many symptoms may be observed. Skin, musculoskeletal, hematologic, and serological involvement are most commonly observed. Some patients show predominately hematologic, renal, or central nervous system manifestations.

Studies have reported that juvenile-onset SLE patients tend to have a more aggressive presentation and course, with higher rates of organ involvement and lower life expectancy than adult-onset SLE patients. Late-onset SLE patients tend to have a more insidious onset of disease and tend to have less major organ involvement and more benign disease course. However, they have a poorer prognosis than patients who developed SLE before the age of 50 years, because of the generally higher frequency of comorbid diseases and higher organ damage, due to aging and longer exposure to ''classical'' vascular risk factors.

Aims of the Study:

To compare clinical and serological differences among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients in our hospital.

DETAILED DESCRIPTION:
Methods:

All patients will be subjected to the following:

1. Thorough medical history of the patients
2. Full clinical examination including:

   1. General examination and vital signs.
   2. Complete rheumatological examination.
   3. SLE disease activity index SLEDAI (ref).
   4. SLICC damage index (ref).
3. Routine investigations (complete blood picture, erythrocyte sedimentation rate and liver functions).
4. Renal investigations:

   1. Kidney functions
   2. Urine analysis
   3. 24 hours protein in urine and/or A/C ratio
   4. Renal biopsy if indicated.
5. ANA test.
6. ANA profile for the most common 19 autoantibodies by immunoblot.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Patients diagnosed as SLE( Systemic lupus erythematosus )according to EULAR / ACE (European League Against Rheumatism /American College of Rheumatology )
2. Age juvenile SLE ( Systemic lupus erythematosus )was defined as a diagnosis below the age of 18 years, and those diagnosed between 19 and 50 years of age were classified as adult SLE ( Systemic lupus erythematosus ), late onset SLE was defined as a diagnosis at more than 50 years of age).
3. Patients with a disease duration of more than 6 months

Exclusion Criteria:

* Exclusion criteria:

  1. Patients with had other autoimmune diseases, such as rheumatoid arthritis, systemic sclerosis, mixed connective tissue disease , overlap syndrome or primary Sjogren's syndrome ,but not secondary Sjogren's syndrome or secondary antiphospholipid syndrome .
  2. Patients who are not willing to be involved in the study

Ages: 6 Months to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 2. Age juvenile SLE was defined as a diagnosis below the age of 18 years, and those diagnosed between 19 and 50 years of age were classified as adult SLE, late onset SLE was defined as a diagnosis at more than 50 years of age).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
serological differences among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients in our hospital. | 1-1-2024
  1. SLE disease activity index SLEDAI (ref) to assessment disease activity in patient .
  2. ANA test (antinuclear antibodies ) to assessment auto-antibodies in different age grouped
laboratory differences among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients in our hospital. | 1-1-2024
  1. Renal biopsy for assessment kidney damage
  2. urine analysis to detect albumin in urine
  3. liver function to detect liver affection
hematological affection among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients in our hospital. | 1-1-2024
  1. cbc complete blood picture to assessment bone marrow affection
  2. erythrocyte sedimentation rate to detect disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: essam mo aboelfadl, professor, Study Director — sohag

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1 Von Feldt JM. Systemic lupus erythematosus. Recognizing its various presentations. Postgrad Med 1995; 97: 79, 83, 86 passim. 2 Estes D, Christian CL. The natural history of systemic lupus erythematosus by prospective analysis. Medicine (Baltimore) 1971; 50: 85-95. 3 Fessler BJ, Boumpas DT. Severe major organ involvement in systemic lupus erythematosus. Diagnosis and management. Rheum Dis Clin North Am 1995; 21: 81-98. 4 Borchers AT, Naguwa SM, Shoenfeld Y, Gershwin ME. The geoepidemiology of systemic lupus erythematosus. Autoimmun Rev 2010; 9: A277-A287. 5 Ferna´ ndez M, Alarco´ n GS, Calvo-Ale´n J, et al. A multiethnic, multicenter cohort of patients with systemic lupus erythematosus (SLE) as a model for the study of ethnic disparities in SLE. Arthritis Rheum 2007; 57: 576-584. 6 Arbuckle MR, James JA, Dennis GJ, et al. Rapid clinical progression to diagnosis among African-American men with systemic lupus erythematosus. Lupus 2003; 12: 99-106.

DOCUMENTS (1):
  • Study Protocol (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT05724940/Prot_000.pdf